CLINICAL TRIAL: NCT03446846
Title: A Randomized, Double-Blind, Parallel-Group, Placebo Controlled Study to Evaluate the Efficacy and Safety of 2 Fixed Doses (5.0 mg or 2.5 mg) of MIN-117 in Adult Patients With Major Depressive Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of MIN-117 in Adult Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minerva Neurosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIN-117C03
Record Dates: First submitted 2018-02-20; First posted 2018-02-27 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MIN-117
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor also masked.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 5.0 mg MIN-117 (Experimental): MIN-117 5.0 mg (consisting of two 2.5 mg capsules) orally daily for 6 weeks
  Interventions: Drug: MIN-117 5.0 mg
- 2.5 mg MIN-117 (Experimental): MIN-117 2.5 mg (consisting of one 2.5 mg capsule and one placebo capsule) orally daily for 6 weeks
  Interventions: Drug: MIN-117 2.5 mg
- Placebo (Placebo Comparator): Placebo (consisting of two placebo capsules) orally daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MIN-117 5.0 mg — 5.0 mg MIN-117 administered as two MIN-117 2.5 mg capsules as a single dose once daily
  Arms: 5.0 mg MIN-117
Drug: MIN-117 2.5 mg — 2.5 mg MIN-117 administered as one MIN-117 2.5 mg capsule and one Placebo capsule as a single dose once daily
  Arms: 2.5 mg MIN-117
Drug: Placebo — Placebo administered as two Placebo capsules as a single dose once daily
  Arms: Placebo

SUMMARY:
MIN-117C03 is a 6-week, 3-arm, randomized, double-blind, placebo controlled study to investigate the safety and efficacy of MIN-117 in male and female patients with Major Depressive Disorder, aged 18 to 65 years. Approximately 324 patients were to be randomly assigned to 1 of 3 treatment arms, including placebo, 2.5 mg MIN-117, or 5.0 mg MIN-117, in a 2:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to read and understand the consent forms, complete study-related procedures, and communicate with the study staff.
* Participants must have provided written consent to participate in the study and understand that they are free to withdraw from the study at any time.
* Participants must have signed the informed consent form for pharmacogenomic research indicating willingness to participate in the pharmacogenomic component of the study in order to participate in the optional pharmacogenomic component of this study. Refusal to consent for this component does not exclude a participant from participation in the clinical study.
* Participants must be aged 18 to 65 years, inclusive, at Screening (Visit 1).
* Meet Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) criteria for diagnosis of moderate or severe major depression with anxious distress and without psychotic features at Screening based on clinical assessment and on the Structured Clinical Interview for DSM-5 (SCID-5). Their major depressive episode must be deemed "valid" using the Massachusetts General Hospital (MGH) State versus trait; Assessability; Face validity; Ecological validity; and Rule of three Ps [pervasive, persistent, and pathological] (SAFER) criteria interview administered by remote, independent raters.
* Participants must be within a body mass index (BMI) of ≥ 18 to < 35 kg/m2 (BMI = weight (kg)/height(m)2] at Screening (Visit 1).
* Participants have a history of at least one previous episode of depression prior to the current episode.
* Participant must have been treated with an antidepressant administered at an adequate dose and duration in the past for the treatment of Major Depression. An adequate treatment is defined as an antidepressant treatment for at least 4 weeks at at least the minimum therapeutic dose, for any particular antidepressant.
* Current major depressive episode of at least 4 weeks in duration.
* At Screening (Visit 1) and Baseline (Visit 2), participants must have a score ≥ 40 on the patient rated Inventory of Depressive Symptoms self-report (IDS-SR30).
* At Screening (Visit 1) and Baseline (Visit 2), participants must have a score ≥ 18 on Hamilton Anxiety Scale (HAM-A).
* At Screening (Visit 1) and Baseline (Visit 2), participants must have a score ≥ 4 on the investigator-rated Clinical Global Impression of Severity Scale (CGI-S).
* Participants must be outpatients at the time of randomization (Baseline [Day 1]).
* Participants must be in good general health prior to study participation with no clinically relevant abnormalities as assessed by the investigator and determined by: medical history, physical examination, vital signs, blood chemistry, hematology, urinalysis, and electrocardiogram (ECG).
* If female, the participant must:

  1. be post-menopausal, or
  2. have had a hysterectomy or tubal ligation or be otherwise incapable of pregnancy, or
  3. must agree to consistent use of 2 methods of contraception for the duration of the study and until 90 days after the last dose of study medication.
* Female participants of childbearing potential must have a negative serum pregnancy test at Screening (Visit 1) and negative serum and urine pregnancy test at Baseline (Visit 2).

Exclusion Criteria:

* A DSM-5 diagnosis of current (active): panic disorder, obsessive compulsive disorder (OCD), post-traumatic stress disorder (PTSD), anorexia nervosa, or bulimia nervosa.
* History or current diagnosis of a psychotic disorder, bipolar disorder, mental retardation, or borderline personality disorders, mood disorder with postpartum onset, somatoform disorders, fibromyalgia, or idiopathic medical conditions.
* At significant clinical risk for suicidal or violent behavior.
* History of treatment within last 6 months with electroconvulsive therapy (ECT), Vagus Nerve Stimulation (VNS), Deep Brain Stimulation (DBS), or Transcranial Magnetic Stimulation (TMS).
* Potential participant who in the opinion of the investigator should not discontinue, or participate in washout of a prohibited concomitant medication.
* Potential participant who demonstrates a greater than 25% decrease in depressive symptoms as reflected by the IDS-SR30 total score from Screening visit to Baseline visit.
* Active cardiovascular disease (including but not limited to: atrial fibrillation or flutter, second and third-degree atrioventricular heart block, resting supraventricular tachycardia > 100 beats per minute, unstable ischemic heart disease, valvular abnormality, sick sinus syndrome or other condition requiring pacemaker) or diastolic blood pressure > 105 mmHg.
* Any serious, untreated, or unstable illnesses, such as: liver or renal insufficiency.
* Any significant pulmonary, endocrine, or metabolic disturbances.
* Documented disease of the central nervous system that could interfere with the study assessments (including by not limited to: stroke, tumor, multiple sclerosis, Parkinson's disease, Alzheimer's disease, Huntington's disease, seizure disorder requiring current anti-convulsants, traumatic brain injury or trauma, and neurosyphilis.
* Hypothyroidism or hyperthyroidism, unless stabilized by appropriate medication for at least 3 months prior to Screening (a normal thyroid-stimulating hormone [TSH] is required prior to randomization at Baseline).
* Any medical condition that can potentially alter oral enteral absorption (e.g., gastrectomy), metabolism (e.g., liver failure), or excretion (e.g., renal failure) of the study drug.
* History of alcohol or substance use disorders (except nicotine and caffeine) meeting DSM-5 criteria within 1-year prior to Screening visit.
* Positive alcohol and urine drug screen for opiates, cocaine, barbiturates, tetrahydrocannabinol, methadone, tricyclic antidepressants, benzodiazepines, and amphetamine/methamphetamine at Screening or Baseline. Patients with positive testing at Screening due to prescribed benzodiazepines, tricyclic antidepressants, barbiturates or opiates are accepted but must test negative at Baseline.
* Male participants who have pregnant partners.
* Received an experimental drug or used an experimental medical device within 60 days before the planned start of treatment (Day 1) or have participated in 2 or more clinical trials in the previous 2 years.
* QT interval corrected with Fridericia's formula (QTcF) at Screening or Baseline greater than 450 msec for males and 470 msec for females.
* Positive hepatitis B surface antigen, or hepatitis C antibody or Human Immunodeficiency Virus (HIV) 1 and 2 antibodies at Screening.
* Employees of the investigator or study center, when the employee has direct involvement in the proposed study or other studies under the direction of that investigator or study center; also family members of the employee or the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (10):
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Collaborative Neuroscience Network, LLC, Torrance, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Hassman Research Institute, LLC, Berlin, New Jersey
  - Neurobehavioral Research, Inc, Cedarhurst, NY, Cedarhurst, New York
  - Neuro-Behavorial Clinical Research Inc, Canton, Ohio
  - Oregon Center for Clinical Investigations, Portland, Oregon
  - FutureSearch Trials, Dallas, Texas
- Bulgaria (9):
  - Mental Health Centre "Prof. Dr. Ivan-Temkov - Burgas" EOOD Complex Lazur, Burgas
  - "University Multiprofile Hospital for Active Treatment - Dr. Georgi Stranski" EAD, First psychiatric clinic, Pleven
  - UMHAT "Sveti Georgi" EAD - Psychiatry Clinic, Plovdiv
  - Mental Health Center, Ruse, Rousse
  - "Diagnostic-Consultative Center St. Vrach and St. St. Kuzma and Damyan" OOD, Psychiatric office, Sofia
  - "Medical Center Stimul" OOD, Psychiatric office, Sofia
  - MC Intermedika, Sofia
  - MC Sveti Naum, Sofia, Sofia
  - DCC Mladost-M OOD, Varna
- Finland (4):
  - Helsingin Psykiatripalvelu Oy at Mehilainen Clinic, Lääkärikeskus Mehiläinen, Helsinki
  - Oulu Mentalcare Oy, Oulu
  - Satakunnan Psykiatripalvelu Oy at Mehiläinen Pori, Pori
  - Mentoria, Tampere
- Georgia (2):
  - Center for Mental Health and Prevention of Addiction Ltd, Tbilisi
  - Tbilisi Mental Health Center Ltd, Tbilisi
- Department of Psychiatry, Addiction and Medical Psychology, Chisinau, Moldova
- Poland (6):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - Ośrodek Badań Klinicznych - Clinsante S.C., Bydgoszcz
  - Zespół Opieki Zdrowotnej w Chełmnie, Poradnia Zdrowia Psychicznego, Chełmno
  - ISPL, Gdansk
  - NZOZ Syntonia, Pruszcz Gdański
  - Prywatna Klinika Psychiatryczna Inventiva, Tuszyn
- Ukraine (15):
  - Communal Institution "Dnipropetrovsk Regional Clinical Hospital n.a. I.I.Mechnykov", Regional Center of Psychosomatic Disorders based on Psychoneurology, Dnipro
  - Municipal non-Profit enterprise "Carpathian Regional Mental, Ivano-Frankivsk
  - State Institution "Institute of Neurology, Psychiatry and Narcology of NAMS of Ukraine" Department of Neuroses and Borderline States, Kharkiv
  - The Training and Research Medical Complex "The Clinic" otharkiv National Medical University, Kharkiv
  - Municipal non-profit enterprise "Kherson Regional Psychiatric Care Facility", Kherson
  - Municipal Non-Profit Enterprise "Kirovohrad Regional Psychoneurological Hospital of Kirovohrad Regional Council, Kropyvnytskyi
  - Municipal enterprise "Heikiv Psychoneurological Hospital, Dnipropetrovsk Regional Council", Kryvyi Rih
  - Kyiv Clinical Hospital on Railway Transport #1 of the branch "Health Center" of the joint-stock company "Ukrainian Railway", Kyiv
  - Kyiv Regional Medical Incorporation Psychiatry Center of Novel Treatment and Rehabilitation of Psychotic Disorders, Kyiv
  - Municipal Institution of Kyiv Regional Council "Regional Psychiatric and Narcological Medical Association", Kyiv
  - National Military-Medical Clinical Center Main Military, Kyiv
  - Municipal non-profit enterprise of Lviv Regional Council "Lviv Regional Clinical Psychiatric Hospital", Lviv
  - Municipal Non-Profit Enterprise "Odessa Regional Psychiatric Hospital # 2" "of Odessa Regional Council", Odesa
  - Communal enterprise "Poltava Regional Clinical Psychiatric Hospital named O.F. Maltsev Poltava Regional Council", Poltava
  - Municipal non-profit enterprise"Vinnytsya Regional Psychoneurological Hospital named Acad. O.I. Yushchenko of Vinnytsya Regional Council, Vinnytsia

RESULTS

PARTICIPANT FLOW:
Groups:
- 5.0 mg MIN-117: MIN-117 5.0 mg taken as two MIN-117 2.5 mg capsules as a single dose orally once daily.
- 2.5 mg MIN-117: MIN-117 2.5 mg taken as one MIN-117 2.5 mg capsule and one Placebo capsule as a single dose orally once daily.
- Placebo: Placebo taken as two Placebo capsules as a single dose orally once daily.
Period: Overall Study
Arm/Group | 5.0 mg MIN-117 | 2.5 mg MIN-117 | Placebo
Started | 90 | 92 | 178
Completed | 83 | 87 | 162
Not Completed | 7 | 5 | 16

BASELINE CHARACTERISTICS:
Population: One patient was randomized to a particular kit # in the Electronic Data Capture system, however, the site dispensed another kit # instead in error. Consequently, the patient was randomized to placebo but received 5.0 mg MIN-117 and was, therefore, included in the (Intent-to-Treat) ITT population based on the randomized treatment to placebo and in the safety population based on the actual treatment they received (5.0 mg MIN-117).
Groups:
- Total: Total of all reporting groups
Arm/Group | 5.0 mg MIN-117 | 2.5 mg MIN-117 | Placebo | Total
Number analyzed (Participants) | 91 | 92 | 177 | 360
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 91 | 92 | 177 | 360
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (11.5) | 47 (12.7) | 47 (12.5) | 48 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 60 | 136 | 258
  Male | 29 | 32 | 41 | 102
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 11 | 20
  White | 85 | 87 | 165 | 337
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a validated, physician-rated scale designed to measure depression severity and detect changes due to antidepressant treatment. The test consists of 10 items, each scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe conditions. MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts. The test exhibits high inter-rater reliability and its capacity to differentiate between responders and nonresponders to antidepressant treatment has been shown to be comparable to the Hamilton Rating Scale for Depression.
Time Frame: Week 6
Population: ITT population: all randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 5.0 mg MIN-117: MIN-117 5.0 mg taken as two MIN-117 2.5 mg capsules as a single dose once daily.
- 2.5 mg MIN-117: MIN-117 2.5 mg taken as one MIN-117 2.5 mg capsule and one Placebo capsule as a single dose once daily.
- Placebo: Placebo taken as two Placebo capsules as a single dose once daily.
Arm/Group | 5.0 mg MIN-117 | 2.5 mg MIN-117 | Placebo
Number analyzed (Participants) | 70 | 76 | 149
score on a scale | -12 (9.2) | -12 (9.2) | -12 (9.2)

2. Secondary Outcome: Change in Hamilton Anxiety Scale (HAM-A)
Description: Hamilton Anxiety Scale (HAM-A) measures the severity of a participant's anxiety, based on 14 parameters, including anxious mood, tension, fears, insomnia, somatic complaints and behavior at the interview. The subject is asked to rate the gravity of each item using a 5-level scale - from 0 to 4, where 0 being not present and 4 being severe - and afterwards, the results are collated and tabulated to determine the severity of anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-25 mild to moderate severity, 25-30 moderate to severe, and >30 indicates very severe. To implement the HAM-A, the acting clinician proceeds through the 14 items, evaluating each criterion independently in form of the five-point scale described above.
Time Frame: Change from Baseline to the end of Week 6
Population: ITT population: all randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5.0 mg MIN-117 | 2.5 mg MIN-117 | Placebo
Number analyzed (Participants) | 70 | 76 | 149
score on a scale | -12 (8.0) | -11 (9.1) | -11 (8.5)

3. Secondary Outcome: Change in Clinical Global Impression of Severity Scale (CGI-S)
Description: The Clinical Global Impression of Severity (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" which is rated on the following scale: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants. The CGI-S will provide an overall clinician-determined summary measure that takes into account all available information including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function.
Time Frame: Change from Baseline to Week 6
Population: ITT population: all randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5.0 mg MIN-117 | 2.5 mg MIN-117 | Placebo
Number analyzed (Participants) | 70 | 76 | 149
score on a scale | -1 (1.3) | -1 (1.1) | -1 (1.2)

4. Secondary Outcome: Change in Clinical Global Impression of Improvement Scale (CGI-I) at Week 6
Description: The Clinical Global Impression of Improvement Scale (CGI-I) will provide an overall clinician-determined summary measure that takes into account all available information including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-I consists of a 7-point scale that evaluates the change from initiation of treatment similar to the Clinical Global Impression of Severity Scale (CGI-S). This 7-point scale requires the clinician to assess how much the subject's illness has improved or worsened relative to a Baseline state at the beginning of the intervention and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: Week 6
Population: ITT population: all randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5.0 mg MIN-117 | 2.5 mg MIN-117 | Placebo
Number analyzed (Participants) | 70 | 76 | 149
score on a scale | 3 (1.0) | 3 (1.2) | 3 (1.1)

ADVERSE EVENTS:
Time Frame: Approximately up to 11 weeks
Description: The Safety Population is the population of all patients who receive at least 1 dose of study treatment. Patients in this population will be analyzed according to the treatment they received, regardless of which treatment they were randomly assigned. All safety and tolerability analyses will be based on this population and treatment assignment. Treatment-emergent adverse events were those that were reported on or after the initiation of the study drug.
Arm/Group | 5.0 mg MIN-117 | 2.5 mg MIN-117 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/92 | 0/177
Serious Adverse Events (participants affected / at risk) | 0/91 | 1/92 | 0/177
Other Adverse Events (participants affected / at risk) | 11/91 | 11/92 | 13/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5.0 mg MIN-117 (N=91) | 2.5 mg MIN-117 (N=92) | Placebo (N=177)
Feeling guilty (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5.0 mg MIN-117 (N=91) | 2.5 mg MIN-117 (N=92) | Placebo (N=177)
Headache (Nervous system disorders) | 11 | 11 | 13

LIMITATIONS AND CAVEATS:
No notable study limitations were identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees not to independently publish the results before the publication of the multi-center results. PI agrees to submit their proposed publication or presentation to Sponsor at least 2 months prior to disclosure. Sponsor may comment and may require deletion of trade secrets and proprietary or confidential information, other than study data.

DOCUMENTS (2):
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT03446846/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT03446846/SAP_001.pdf